CLINICAL TRIAL: NCT02343575
Title: Valproic Acid for Treatment of Hyperactive or Mixed Delirium in ICU
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We did not recruit the research assistant and terminated the study
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yelizaveta Sher, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28330
Record Dates: First submitted 2015-01-08; First posted 2015-01-22 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Hyperactive Delirium; Mixed Delirium
Keywords: Hyperactive delirium; Mixed delirium; Anti-psychotic; Haldol; Valproic Acid
MeSH Terms: interventions — Valproic Acid; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valproic Acid (Experimental): 1. Start:
     VPA PO/NGT 500 mg BID
  2. If need to increase in 24 or more hours:
     VPA 500 mg PO/NGT q am, 1000 mg PO/NGT QHS
  3. If need to increase in 24 or more hours:
     VPA 500 mg PO/NGT q am, 1500 mg PO/NGT QHS
  4. If need to increase in 24 or more hours:
  VPA 500 mg PO/NGT Q am, 2000 mg PO/NGT QHS
  Rescue at all stages: HAL IV 2-5 mg Q4hr PRN
  Interventions: Drug: Valproic Acid; Drug: Haloperidol
- Placebo (Placebo Comparator): Placebo: PO/NGT BID
  Rescue: HAL IV 2-5 mg Q4hr PRN
  Interventions: Drug: Placebo; Drug: Haloperidol

INTERVENTIONS:
Drug: Valproic Acid — 1.
  Start:
  VPA PO/NGT 500 mg BID
  2.
  If need to increase in 24 or more hours:
  VPA 500 mg PO/NGT q am, 1000 mg PO/NGT QHS
  3.
  If need to increase in 24 or more hours:
  VPA 500 mg PO/NGT q am, 1500 mg PO/NGT QHS
  4.If need to increase in 24 or more hours:
  VPA 500 mg PO/NGT Q am, 2000 mg PO/NGT QHS
  Other Names: VPA; Valproate; Depakote
  Arms: Valproic Acid
Drug: Placebo — Placebo 500 mg matched to VPA BID PO/NGT
  Arms: Placebo
Drug: Haloperidol — Both arms (intervention VPA and placebo) will receive flexible as needed haloperidol: Rescue: HAL IV 2-5 mg Q4hr PRN
  Other Names: Haldol

SUMMARY:
Delirium is the most often encountered psychiatric diagnosis in the general hospital, with incidence up to 85% in the intensive care unit (ICU) setting and with significant consequences on patients' morbidity and mortality. Currently, although not FDA approved, antipsychotics are often considered the first-line pharmacological treatment. However, there can be limitations to their use, including side effects or lack of efficacy. Valproic acid (VPA) is one of the alternatives at times used in such patients which from limited case series data appears to be helpful and tolerated. VPA can provide relief from agitation that poses a threat to the safety and recovery of the patient. Moreover, mechanistically it addresses the neurochemical and cellular abnormalities inherent in delirium (it has NMDA-antagonist, anti-dopaminergic, GABAergic,anti-inflammatory, anti-apoptotic, and histone deacetylase inhibitor properties, among others). The purpose of this study is to evaluate the efficacy and tolerability of the VPA in the first known to us randomized controlled trial.

DETAILED DESCRIPTION:
The investigators plan to investigate the efficacy and tolerability of scheduled VPA as compared to placebo with as needed basis (PRN) haloperidol (as a back-up in both arms) for treatment of hyperactive or mixed delirium. Patients will be randomized to scheduled VPA or placebo (normal saline) and both arms will have flexible PRN dosing of haloperidol. Thus, the investigators plan to learn the time to delirium resolution in patients treated with VPA versus placebo; percentage of patients responding to VPA versus placebo; tolerability of VPA versus placebo. If addition of scheduled VPA proves to shorten time to delirium resolution as compared to placebo, lead to less use of haloperidol, and/or have fewer side effects, it would provide a very important addition to our limited evidence-based repertoire of delirium treatment. Moreover, this pilot study would then pave the way for the bigger randomized control trial powered to detect its effect size.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age and older
* admitted to surgical ICU
* diagnosed with hyperactive or mixed delirium

Exclusion Criteria:

* hypoactive delirium
* primary team does not think patient is appropriate to participate
* no oral access (PO or NGT)
* non-English speaking
* contraindication to study medications
* pregnant women or woman of child-bearing age not on documented contraception
* QTc = or greater than 480
* hepatic dysfunction
* decreased platelets or platelet dysfunction
* bleeding disorder, current major bleeding
* history of NMS, epilepsy, or PD
* diagnosis of schizophrenia, bipolar disorder or schizoaffective disorder
* on warfarin or carbapenems
* delirium due to alcohol withdrawal
* treated with antipsychotics for more than 48 hours prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelizaveta Sher, M.D., Principal Investigator — Stanford University; Jose R Maldonado, M.D., Study Director — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Valproic Acid: Participants received Valproic Acid (VPA) and flexible haloperidol as needed.
- Placebo: Participants received VPA placebo and flexible haloperidol as needed.
Period: Overall Study
Arm/Group | Valproic Acid | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Valproic Acid: Participants received VPA and flexible haloperidol as needed.
- Total: Total of all reporting groups
Arm/Group | Valproic Acid | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Delirium Resolution
Description: Delirium resolution was defined as three negative Confusion Assessment Method (CAM) assessments, performed by nurses every 12 hours.
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 1 | 2
days | 2 | 1.5 (0.7)

2. Secondary Outcome: Use of as Needed Anti-psychotic Agent
Description: Amount of Haldol administered.
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 1 | 2
mg | 0 | 1 (1.2)

3. Secondary Outcome: Side Effects From Medications
Description: Side effects may have included liver function test (LFT) increase, platelet decrease, bleeding, or QTc prolongation.
Time Frame: Up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 1 | 2
Participants
  LFT increase | 0 | 0
  Platelet decrease | 0 | 0
  Bleeding | 0 | 0
  QTc prolongation | 0 | 1

4. Secondary Outcome: Intensity of Delirium as Measured by the Intensive Care Delirium Screening Checklist (ICDSC) Delirium Severity Scale
Description: The items include the assessment of: (1) consciousness ( deep sedation/coma, agitation, normal wakefulness, or light sedation); (2) inattention; (3) disorientation; (4) hallucination, delusion, or psychosis; (5) psychomotor agitation or retardation; (6) inappropriate speech or mood; (7) sleep-wake cycle disturbances; and (8) fluctuation of symptomatology. The maximum score is eight; scores of ≥4 indicate the presence of delirium and score zero is indicate not in delirium. Each item is scored 0-8.
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | 5 | 4 (2.7)

5. Secondary Outcome: Length of ICU Stay
Time Frame: During expected average hospitalization (of 1 month)
Population: Data were not collected for this outcome
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Length of Hospital Stay
Description: Participation in the study ended once delirium was resolved and the patient was off study drug. This outcome presents the total length of hospital stay, which may have been longer than participation in the study.
Time Frame: During expected average hospitalization (of 1 month)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 1 | 2
days | 4 | 8 (8.5)

ADVERSE EVENTS:
Time Frame: Up to 5 days
Arm/Group | Valproic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valproic Acid (N=1) | Placebo (N=2)
QTc prolongation (Cardiac disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study terminated early and did not meet its planned sample size of 30 participants, leading to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-03-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT02343575/Prot_000.pdf